CLINICAL TRIAL: NCT06097572
Title: Improved Diagnostics in Food Allergy (ID-in-FA) Study
Brief Title: Improved Diagnostics in Food Allergy Study
Acronym: ID-in-FA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal College of Surgeons, Ireland (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22SM7832; 22/NW/0321 (Other: NHS Human Research Authority)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut (Experimental): Participants with possible allergy to peanut
  Interventions: Diagnostic Test: Intranasal food challenge; Diagnostic Test: Mast cell activation test
- Cow's Milk (Experimental): Participants with possible allergy to cow's milk
  Interventions: Diagnostic Test: Intranasal food challenge; Diagnostic Test: Mast cell activation test

INTERVENTIONS:
Diagnostic Test: Intranasal food challenge — Subjects will undergo an incremental intranasal challenge to initially 0.9% NaCl saline solution, and then increasing doses of the food protein
Diagnostic Test: Mast cell activation test — Blood will be processed for mast cell activation as previously described (https://doi.org/10.1016/j.jaci.2018.01.043)

SUMMARY:
The investigators will conduct low-dose intranasal allergen challenges on children and young people with an indeterminate diagnosis of food allergy to cow's milk or peanut. Blood samples will also be taken, for conventional blood allergy diagnostics (allergy-specific Immunoglobulin E) and mast cell activation test (MAT). The data will be used to determine the diagnostic accuracy of two complementary, novel approaches to diagnose food allergy, in a representative clinical cohort.

ELIGIBILITY:
Inclusion Criteria:

* IgE-sensitisation to peanut, (hen's) egg or cow's milk, with indeterminate clinical (allergy) status, defined as IgE-sensitisation below 95% positive predictive value (PPV) for diagnosis for either allergen-specific IgE or SPT, using published cut-offs OR clinician suspicion of tolerance (on basis of clinical history) despite IgE sensitisation >95% PPV cut-offs.
* Written informed consent from parent/guardian, with assent from children aged 6 years and above wherever possible. Participants aged over 16 years will need to provide their own informed consent.

Exclusion Criteria:

* Acute illness or current unstable asthma, defined as:

  1. Febrile ≥38.0oC in last 72 hours
  2. Acute wheeze in last 72 hours requiring treatment
  3. Recent admission to hospital in preceding 2 weeks for acute asthma
* Current medication

  1. Asthma reliever medication required in preceding 72 hours
  2. Recent administration of a medicine containing antihistamine within the last 3 days
  3. Current oral steroid for asthma exacerbation or course completed within last 2 weeks
* Unwilling or unable to fulfil study requirements

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Test performance | 1 day
  Comparison of test performance characteristics (sensitivity, specificity, measured according to standard statistical methods) for each of the following diagnostic tests, compared to a formal oral food challenge (FC) as the reference standard:
  i. Intranasal FC (InFC) ii. Skin prick testing iii. Characterisation of serum-specific IgE to whole allergen, components and molecular components iv. Mast cell activation test (MAT) v. Basophil activation test (BAT) (peanut only)

SECONDARY OUTCOMES:
Adverse events | 1 day
  Number of participants who experience a non-allergic adverse event, and/or have symptoms of a systemic allergic reaction) associated with the intranasal food challenge.

CONTACTS AND LOCATIONS:
Locations (2):
- Prof Jonathan Hourihane, Dublin, Ireland
- Imperial College Healthcare NHS Trust (St. Mary's Hospital), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared upon request to the Chief Investigator.